CLINICAL TRIAL: NCT01864343
Title: Target Temperature Management In Myocardial Infarction - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christoph Testori, Department of Emergency Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STATIM-Pilot; MUW_492/2011
Record Dates: First submitted 2013-05-17; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Myocardial Infarction; Myocardial Reperfusion Injury; Reperfusion Injury; Anterior Wall Myocardial Infarction; Inferior Wall Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Myocardial Reperfusion Injury; Reperfusion Injury; Anterior Wall Myocardial Infarction; Inferior Wall Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre- and perinterventional hypothermia (Experimental): Cooling will be initiated by the application of cooling pads in the out-of-hospital setting followed by an infusion of 1000-2000ml of cold saline. In the cath lab a endovascular cooling catheter will be placed into the inferior vena cava via a femoral vein to achieve a core temperature of <35°C prior to revascularization.
  Interventions: Device: EMCOOLS flex pad; Philips Innercool RTx

INTERVENTIONS:
Device: EMCOOLS flex pad; Philips Innercool RTx — Surface cooling with EMCOOLS flex pads (out-of-hospital); Infusion of 1000ml to 2000ml of cold saline (out-of-hospital); central-venous cooling (Philips Innercool RTx)

SUMMARY:
The primary goal in the treatment of acute myocardial infarction is to reperfuse the ischemic myocardium to reduce infarct size. Animal data and human data suggest that whole-body cooling to temperatures below 35°C before revascularisation can additionally reduce infarct size and therefore improves outcome in these patients.

The purpose of the study is to determine the feasibility and safety of a combined cooling strategy started in the out-of-hospital arena for achieving pre-reperfusion hypothermia in patients with acute st-elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Immediately transfer to cath-lab is possible
* Anterior or inferior ST-Elevation myocardial infarction
* ST-Segment elevation of >0.2mV in 2 or more anatomically contiguous leads
* Duration of symptoms <6 hours

Exclusion Criteria:

* Participation in another study
* Patients presenting with cardiac arrest
* Tympanic temperature of <35.0°C prior enrolment
* Thrombolysis therapy
* Previous myocardial infarction in medical history
* Previous percutaneous coronary intervention or coronary artery bypass graft
* Severe heart failure (defined as a New York Heart Association (NYHA) score of III or IV), Killip class II through IV at presentation
* Clinical signs of infection
* End-stage kidney disease or hepatic failure
* Recent stroke (within the last six month)
* Conditions that may be exacerbated by hypothermia, such as haematological dyscrasias, oral anticoagulant treatment with international normalized radio >1.5, severe pulmonary disease
* Pregnancy. Women of childbearing potential are excluded
* Allergy to meperidine, buspirone, magnesium, or polyvinyl chloride
* Use of a monoamine oxidase inhibitor such as selegiline in the previous 14 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of a combined cooling strategy for achieving a core temperature of <35.0°C at the time of reperfusion of the infarct related artery | Time of reperfusion of the culprit lesion in st-elevation myocardial infarction (expected average 120 minutes)
  Blood temperature will be recorded at the time of first wire-crossed lesion of the infarct related coronary stenosis

SECONDARY OUTCOMES:
Safety of a combined cooling strategy as an adjunctive therapy on primary percutaneous coronary intervention in acute st-elevation myocardial infarction | within 45 days (+/- 15 days)
  Incidence of major adverse cardiac events as defined as: death, heart failure, pulmonary edema, recurrent MI, malignant arrhythmias (i.e. ventricular fibrillation, sustained ventricular tachycardia) emergent stent revascularisation, any hospitalisation, major/minor bleeding (according to TIMI-bleeding score), infection (clinical relevant infection with the need of systemic antimicrobiotic therapy) within a period of 45±15 days
Tolerability of a combined cooling strategy as an adjunctive therapy on primary percutaneous coronary intervention in acute st-elevation myocardial infarction | during active cooling and rewarming (in average the first 4 hours)
  Patients are monitored for incidence of shivering using a 4-point scale: 0, no shivering evident; 1, isolated facial or masticatory fasciculation; 2, peripheral shivering; 3, uncontrolled rigor during the cooling procedure (in average the first 4 hours)
Time to revascularisation (first medical contact to balloon time) | Time of reperfusion (in average 120 minutes)
  The time to reperfusion of the infarct related artery is crucial in acute ST-elevation myocardial infarction. To evaluate if the cooling procedure has a substantial influence on this time frame we measure the time from first medical contact to reperfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Testori, MD, Principal Investigator — Medical University of Vienna, Dept. of Emergency Medicine
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Testori C, Sterz F, Delle-Karth G, Malzer R, Holzer M, Stratil P, Stockl M, Weiser C, van Tulder R, Gangl C, Sebald D, Zajicek A, Buchinger A, Lang I. Strategic target temperature management in myocardial infarction--a feasibility trial. Heart. 2013 Nov;99(22):1663-7. doi: 10.1136/heartjnl-2013-304624. Epub 2013 Sep 24. PMID 24064228